CLINICAL TRIAL: NCT03043469
Title: Dysfunctional Breathing: Multidimensional Characterisation and Assessment Tool
Brief Title: Dysfunctional Breathing: Characterisation and Assessment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Brunel University (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Lais Silva Vidotto, Ms Lais Silva Vidotto, Brunel University
Other Study IDs: 1468-NHS-Dec/2016- 4775-1
Record Dates: First submitted 2017-01-30; First posted 2017-02-06 (Estimated); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Respiration Disorder; Hyperventilation Syndrome; Breathlessness; Breath Shortness
Keywords: dysfunctional breathing
MeSH Terms: conditions — Respiration Disorders; Dyspnea | interventions — Demography; Body Height; Weights and Measures; Aging; Sex; 4-amino-4'-hydroxylaminodiphenylsulfone; Patient Health Questionnaire; Exercise Test; Calorimetry, Indirect; Respiratory Function Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy participants: Day 1: Hospital assessments (~3 hours): Demographic data, Manual Assessment of Respiratory Motion, Slow-breathing task, Six-minute exercise test, Indirect calorimetry, Oxygen saturation monitoring, heart rate variability analysis, continuous measurement of arterial blood pressure, lung function test, the Nijmegen Questionnaire and the Self-Evaluation of Breathing Questionnaire, the Hospital anxiety and depression scale, and the Short-Form Survey Instrument, Breath-hold test, Lung function test, respiratory muscle function assessment.
  Days 2-8: Physical Activity Monitoring
  Interventions: Other: Short-form survey instrument; Other: Demographic data; Other: Hospital Anxiety and Depression Scale; Other: Nijmegen questionnaire; Other: The Self-evaluation of breathing questionnaire; Other: six-minute exercise test; Other: Indirect calorimetry; Other: Oxygen saturation monitoring; Other: Heart rate variability analysis; Other: Continuous measurement of arterial blood pressure; Diagnostic Test: Lung function test; Other: Respiratory muscle function; Other: Manual assessment of respiratory motion; Other: Breath-hold test; Other: Physical Activity monitoring
- Restrictive lung disease group: Day 1: Hospital assessments (~3 hours): Demographic data, Manual Assessment of Respiratory Motion, Slow-breathing task, Six-minute exercise test, Indirect calorimetry, Oxygen saturation monitoring, heart rate variability analysis, continuous measurement of arterial blood pressure, lung function test, the Nijmegen Questionnaire and the Self-Evaluation of Breathing Questionnaire, the Hospital anxiety and depression scale, and the Short-Form Survey Instrument, Breath-hold test, Lung function test, respiratory muscle function assessment.
  Days 2-8: Physical Activity Monitoring
  Interventions: Other: Short-form survey instrument; Other: Demographic data; Other: Hospital Anxiety and Depression Scale; Other: Nijmegen questionnaire; Other: The Self-evaluation of breathing questionnaire; Other: six-minute exercise test; Other: Indirect calorimetry; Other: Oxygen saturation monitoring; Other: Heart rate variability analysis; Other: Continuous measurement of arterial blood pressure; Diagnostic Test: Lung function test; Other: Respiratory muscle function; Other: Manual assessment of respiratory motion; Other: Breath-hold test; Other: Physical Activity monitoring
- Primary dysfunctional Breathing group: Day 1: Hospital assessments (~3 hours): Demographic data, Manual Assessment of Respiratory Motion, Slow-breathing task, Six-minute exercise test, Indirect calorimetry, Oxygen saturation monitoring, heart rate variability analysis, continuous measurement of arterial blood pressure, lung function test, the Nijmegen Questionnaire and the Self-Evaluation of Breathing Questionnaire, the Hospital anxiety and depression scale, and the Short-Form Survey Instrument, Breath-hold test, Lung function test, respiratory muscle function assessment.
  Days 2-8: Physical Activity Monitoring
  Interventions: Other: Short-form survey instrument; Other: Demographic data; Other: Hospital Anxiety and Depression Scale; Other: Nijmegen questionnaire; Other: The Self-evaluation of breathing questionnaire; Other: six-minute exercise test; Other: Indirect calorimetry; Other: Oxygen saturation monitoring; Other: Heart rate variability analysis; Other: Continuous measurement of arterial blood pressure; Diagnostic Test: Lung function test; Other: Respiratory muscle function; Other: Manual assessment of respiratory motion; Other: Breath-hold test; Other: Physical Activity monitoring
- Secondary dysfunctional breathing group: Day 1: Hospital assessments (~3 hours): Demographic data, Manual Assessment of Respiratory Motion, Slow-breathing task, Six-minute exercise test, Indirect calorimetry, Oxygen saturation monitoring, heart rate variability analysis, continuous measurement of arterial blood pressure, lung function test, the Nijmegen Questionnaire and the Self-Evaluation of Breathing Questionnaire, the Hospital anxiety and depression scale, Asthma Control Questionnaire, and the Short-Form Survey Instrument, Breath-hold test, Lung function test, respiratory muscle function assessment.
  Days 2-8: Physical Activity Monitoring
  Interventions: Other: Short-form survey instrument; Other: Demographic data; Other: Hospital Anxiety and Depression Scale; Other: Nijmegen questionnaire; Other: The Self-evaluation of breathing questionnaire; Other: six-minute exercise test; Other: Indirect calorimetry; Other: Oxygen saturation monitoring; Other: Heart rate variability analysis; Other: Continuous measurement of arterial blood pressure; Diagnostic Test: Lung function test; Other: Respiratory muscle function; Other: Manual assessment of respiratory motion; Other: Breath-hold test; Other: Physical Activity monitoring; Other: Asthma Control Questionnaire

INTERVENTIONS:
Other: Short-form survey instrument — Questionnaire with questions about quality of life. Takes about 5 minutes to be completed.
  Other Names: SF-36
Other: Demographic data — height, weight, age, gender, list of comorbidities, health history, level of physical activity, medicines in use. Takes about 10 minutes to be completed.
  Other Names: height, weight, age, gender
Other: Hospital Anxiety and Depression Scale — Questionnaire with questions about anxiety and depression. Takes about 5 minutes to be completed.
  Other Names: anxiety and depression questionnaire
Other: Nijmegen questionnaire — Answering questions about symptoms related to breathing. Takes about 5 minutes to be completed.
Other: The Self-evaluation of breathing questionnaire — Answering questions about self-evaluation of breathing. Takes about 5 minutes to be completed
Other: six-minute exercise test — Cycling against certain load in a bicycle for 6 minutes. Takes about 16 minutes to be completed together with indirect calorimetry, oxygen saturation monitoring, heart rate variability analysis and continuous monitoring of arterial blood pressure).
Other: Indirect calorimetry — Breathing through a mask that measures levels of oxygen, carbon dioxide, breathing frequency and others (non-invasively). Takes about 16 minutes to be completed, together with the 6-minute exercise test.
  Other Names: gas analysis
Other: Oxygen saturation monitoring — The measurement of the amount of oxygen which is attached to haemoglobin molecules (non-invasively). Takes about 16 minutes to be completed, together with the 6-minute exercise test.
Other: Heart rate variability analysis — Measurement of the variation in the beat-to-beat interval (non-invasively). Takes about 16 minutes to be completed, together with the 6-minute exercise test.
Other: Continuous measurement of arterial blood pressure — Measurement of blood pressure based on the peripheral pulse using a finger cuff (non-invasively). Takes about 16 minutes to be completed, together with the 6-minute exercise test.
Diagnostic Test: Lung function test — Breathing through a mouth-piece in many different ways in order to measure the function of the lungs (non-invasively).
Other: Respiratory muscle function — Breathing through a mouth-piece in many different ways in order to measure the function of the respiratory muscles (non-invasively).
Other: Manual assessment of respiratory motion — Measure of the movements of the thorax while the participant is breathing (non-invasively).
Other: Breath-hold test — Holding the breath a few times for as long as possible.
Other: Physical Activity monitoring — Wearing a light-weight activity monitor to be wore on the hip for 7 consecutive days during, at least, 8 hours per day.
Other: Asthma Control Questionnaire — Only for asthmatics: answering questions about the control the participant has over this respiratory condition/symptoms.
  Groups: Secondary dysfunctional breathing group

SUMMARY:
Dysfunctional breathing (DB) is a respiratory condition characterised by an abnormal breathing pattern, among other complaints, that can occur either in the absence of other pathophysiology (primary DB), e.g. anxiety-related factors, or secondary to cardiopulmonary disease (secondary DB), e.g. asthma. As a consequence, patients may experience breathlessness and present with periods of increased ventilation or erratic breathing, interspersed with episodes of breath holding or deep sighs. In addition to respiratory symptoms, DB also generates non- respiratory symptoms (e.g. dizziness and increased heart rate). It is estimated 1 in 10 people in the United Kingdom (UK) have DB. However, DB remains poorly understood, with no standardised approach to diagnosis and assessment.

The purposes of this study are:

Study 1) To identify physiological, functional and psychological characteristics of participants with DB compared to healthy participants.

Firstly, symptoms, lung function, respiratory gas analysis, exercise capacity, respiratory muscle function, respiratory motion, level of physical activity, quality of life and anxiety & depression scores will be assessed in 20 participants with primary DB, 20 with secondary DB and compared to 20 healthy participants.

Study 2) To develop an assessment tool based on physiological, functional or psychological variables found to be different between any of the 3 groups in Study 1.

In order to do that, 54 people with DB (between primary and secondary) and 27 people presenting with breathlessness secondary to restrictive lung disease will be assessed. Analysis of these data will determine whether these variables can be used as a diagnostic tool capable of distinguishing DB from restrictive lung diseases characterised by breathlessness.

The recruitment period will be 1-2 years, with an individual participation of 9 days; 1-day on site testing, plus 7-day home activity monitoring, and 1 day to return the activity monitor (which will happen whenever the participant needs to return to the site).

DETAILED DESCRIPTION:
In this research, the aims are: 1) to characterise and compare participants with primary dysfunctional breathing (DB), secondary DB and healthy participants, 2) to develop an assessment and identification tool for the population with DB, 3) to identify subgroups of people with DB based on their functional, physiological and psychological characteristics.

In order to do that, in Study 1, there will be a comparison of many different aspects (described below) between three groups of 20 participants each: primary DB, secondary DB and healthy participants. With the results of these comparisons, it will be possible to know more about the differences people with DB have in relation to the healthy population, and to describe their main characteristics. Based on that, in Study 2, it will be possible to select the variables that are different between groups and replicate those tests in an extra 54 participants DB (primary and secondary) and 27 with breathlessness secondary to restrictive lung disease (DB excluded). The second stage will suggest tests to be used when identifying and evaluating this population, and statistically identify subgroups of people with DB based on their characteristics.

It is important to note why the inclusion of healthy participants and participants with breathlessness secondary to restrictive lung disease is important in this research programme. Firstly, it is essential to know the main characteristics of DB in relation to the healthy population. Secondly, the assessment tool has to be able to suggest probability of negative diagnosis of DB for people who do not have DB, and not only positive diagnosis for those who have.

There are no standardised criteria available to diagnose DB. However, experienced chest physicians at Guy's and St Thomas' Foundation Trust (GSTFT) identify probable DB, and provide a clinical diagnosis (CD) according to the following criteria: patients presenting with symptoms that are not concordant with the severity of the underlying health condition (in case of secondary DB), patients presenting with symptoms that persist despite optimal disease management and/or no objective markers of deterioration/exacerbation (in case of secondary DB), patients presenting with symptoms in the presence of negative tests for organic cause/medically unexplained (in case of primary DB), patients presenting with symptoms that are considered functional (in case of primary DB).

Ability to comprehend and/or perform the procedures of this research, as well as the presence of major orthopaedic, neurological or cardiac conditions will be checked by Leyla Osman and the Chest physicians via medical records and when the possible participant is approached to receive information about the study. For example: health conditions in which patients present with an impairment of mental faculties and/or motor function (inability to cycle with no discomfort).

Healthy participants will be contacted via email list at Brunel University London, and via flyers placed on the University's and Hospital's website and murals (attached). Participants with restrictive lung disease will be reached in person or via telephone call when they are referred to respiratory physiotherapy, or via flyers placed on the Hospital's murals. Because there are not plenty of patients with DB, those who are already registered on the Hospital's system as presenting with DB (assessed by a chest physician) will be called. New patients with DB will be contacted in person or via telephone call by the respiratory physiotherapist of the clinical team (Leyla Osman).

If those contacted about this research are interested in taking part in this study, they will be provided with the participant information sheet, have the opportunity to ask any questions they may have and it will be checked if they meet the inclusion criteria. Before starting the assessments, they will be asked to sign the informed consent.

When signing the informed consent, participants will be asked a few questions:

Please, tick this box if you authorise the researchers of this study to have access to your medical records Please, tick this box if you are aware that your General practitioner will be informed about your participation in this research Please, tick this box if you would like to receive a report with your results of the tests performed in this study (within 30 days from the end of your assessments) Please, tick this box if you would like us to contact you in the future to inform you about the final results of this study Please, tick this box if you are participating in other study/ies at this moment. If yes, please mention below what this/these study/ies is/are about and the contact of the person responsible for it The assessments will be performed by Lais Silva Vidotto (respiratory physiotherapist and researcher) at the Hospital/University over a period of approximately 3 hours. Many of these assessments form part of routine hospital investigations for patients with DB. Duration may vary depending on individual needs and limitations, such as time given to recover from any physical or mental effort. Secondly, a physical activity monitor will be given to all participants, which will be returned to the researchers on the next medical appointment at the Hospital/classes at the University (classes at the University in case of healthy participants). During the 3-hour assessment they will have the opportunity to rest whenever is necessary and snacks and refreshments will be provided in the intervals (caffeine-free ingredients).

Assessments and their approximate duration are as follows: demographic information (10 minutes), health-related quality of life questionnaire (SF-36) (5 minutes), Hospital anxiety and depression scale (HADS) (5 minutes), Nijmegen questionnaire (NQ) (5 minutes), Self-evaluation of breathing questionnaire (SEBQ) (5 minutes), Asthma Questionnaire (only for asthmatics) (5 minutes), lung function test (30 minutes), respiratory muscle function (30 minutes, assessment of the respiratory movements (MARM) (10 minutes), breath-hold test (BHT) (20 minutes), slow-breathing task (15 minutes) and the sub-maximal exercise test (10 minutes) (during the two last tests participants will be wearing small and light-weight devices that monitor heart activity, breathing function and blood pressure and take 15 minutes to be placed all together).

Day 1: Hospital assessments (~3 hours) The tests will be performed in a private room at St Thomas' Hospital or Brunel University London. Participants will be advised to stay 48 hours without practicing exercise. Also, they will be instructed to take all the medicines they normally use and to report their names and doses to the examiner.

1. Patients will be asked about their medical history, date of birth and symptoms. Also, participants' weight and height will be measured.
2. Chest movements while breathing:

   At this stage, participants are going to stand still while the researcher will place their hands on the back of their chests in order to evaluate its movements while participants are breathing. This is going to take about 10 minutes.
3. Slow-breathing task:

   Participants will be instructed on how to breathe slower (6-10 bpm) for a few minutes (5-15 minutes) and will keep wearing the mask, the heart rate monitor and the arterial blood pressure monitor during this task.
4. Exercise test, breathing and cardiovascular function:

   Light-weight devices will be attached to participants' chest (cardiac monitor), in order to evaluate heart function, to their faces (mask-gas analyser) to assess respiratory function, and to their non-dominant arm (arm and finger), to assess blood pressure. The device used to assess blood pressure continuously measures the pulse of the finger, calibrated by an arm cuff, with no discomfort to the participant. Those assessments will be performed while participants rest for five minutes, while they cycle on a bicycle with moderate resistance for six minutes, and while they rest for five more minutes. Just before the exercise test, at the third minute, and just after it, participants will be asked about any leg or breathing discomfort and how mindful they are in relation to discomfort related to the task. Approximate time of this task: 16 minutes.
5. Questionnaires:

   Participants will be asked to fill in some questionnaires that will ask about their breathing and quality of life and will take about 25 minutes to complete. Participants will be asked to complete these questionnaires after having the opportunity to ask questions about them.
6. Breath hold test:

   Participants will be asked to hold their breath for as long as they can for 3 times, resting for 5 minutes after each one of them, and the researcher will use a stopwatch in order to count the time they are able to do it. The whole task will last in approximately 20 minutes.
7. Lung and respiratory muscle function assessments:

Researchers will use three devices to measure the function of participants' lungs and respiratory muscles. They will be asked to breathe in and out in several different ways, wearing a nose clip, so that researchers can record their general breathing function. This is going to take about one hour to finish.

At the end of the assessment session, participants will be instructed on how to use a device that measures the level of physical activity.

Days 2-8: Physical Activity Monitoring Participants will be asked to wear two small activity monitors attached to their hip for 7 consecutive days, keeping their routine as normal as possible. Participants will have to use the equipment for at least 8 hours/day while they are awake, excluding water activities (e.g. shower) and sleeping, writing down the exact time they put it on and the time they took this off.

Day 9: Return of the activity monitors Participants recruited from Brunel University London will return their physical activity monitors to the researchers on their next visit to the University (for classes, meetings etc.); those recruited from GSTFT will return it on their next hospital appointment.

Although this study requires a cross-sectional design, it may take a long period to be completed, since patients with DB are not easily identified and referred to other health professionals to receive specific diagnosis or treatment. Considering this difficulty in finding participants with DB, justified by the fact that there is no established way of identifying these patients, this research may take 1-2 years to be completed. However, It will enable the researchers to look at every single result and be rigorous with the quality of the data collected. In order to do that, the researchers will not wait for all assessments to be finished to process and plot the data. Every time a participant is evaluated, their results will be organised and plotted within the next few days. It will also enable the data to be statistically analysed when needed.

ELIGIBILITY:
Inclusion Criteria:

* patients with DB (according to the CD)
* healthy people
* aged 18 or over,
* must be able to comprehend and/or perform the procedures of this research
* must be able to consent to participate
* people with signs of breathlessness secondary to restrictive lung disease (DB excluded)

Exclusion Criteria:

* people whose condition is unstable or have experienced an exacerbation of symptoms over the last 4 weeks
* patients who are oxygen-dependant (at rest or during exercise),
* those who are on oral steroids or have completed a course of those medications less than four weeks prior to the assessment day,
* those who have major orthopaedic, neurological or cardiac conditions
* those who received breathing retraining before

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with primary/secondary dysfunctional breathing and patients with restrictive lung diseases will be recruited from clinics of respiratory medicine (secondary care). Healthy participants will be recruited from the general population (at Brunel University London).
Sampling Method: Non-Probability Sample
Enrollment: 141 (Estimated)
Dates: Start 2020-08-08 (Estimated); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
Signs of Anxiety and Depression | This scale will be applied only once during the first day of assessment and takes about 5 minutes for the participant to complete.
  Anxiety and depression will be evaluated by the widely used Hospital Anxiety and Depression Scale (HADS), developed by Zigmond and Snaith (1983) to identify and screen cases of anxiety and depression in non-psychiatric environments. It has been proven to be a valid psychological instrument (Bjelland et al. 2002). The HADS is subdivided into two subscales with seven questions each: Anxiety (HADS-A) and Depression (HADS-B). Therefore, it is able to differentiate anxiety from depression possible/probable disorders.
Levels of subjective sensation related to Hyperventilation Syndrome | This scale will be applied only once and takes about 5 minutes to be completed by the participant.
  The Nijmegen Questionnaire is a clinically used tool for analysis of 16 symptoms related to Hyperventilation syndrome arising from different body systems (such as chest pain, blurred vision and faster or deeper breathing). The participant will choose the answer from a 5-point ordinal scale considering the frequency of symptoms. 23 of 64 points or more is considered positive for abnormality of subjective sensations (van Dixhoorn and Folgering 2015) and correlates positively with Dysfunctional Breathing (Vansteenkiste, Rochette, Demedt, 1991).
Self-evaluation of breathing | This scale will be applied only once and takes about 5 minutes to be completed by the participant..
  The Self Evaluation Breathing Questionnaire is a reliable tool developed by Courtney and Greenwood (2009) to assess breathing pattern of participants with Dysfunctional Breathing (Mitchell et al. 2015). It contains 17 items that are answered using a 4-point Likert scale and includes two main factors: "lack of air", which is about feeling and sensing; and "perception of inappropriate or restricted breathing", which is about observing or noticing. It has been indicated that the higher the SEBQ score, the more severe is the clinical condition of Dysfunctional Breathing (Mitchell et al. 2015). However, researchers who created the SEBQ questionnaire suggested that it can be used as a screening tool for identifying Dysfunctional Breathing and for monitoring changes in breathing symptoms after treatment, but there is no normal value available in the literature for this questionnaire yet (Courtney, Greenwood, et al. 2011).
Respiratory Motion | This assessment will be applied only once and takes about 10 minutes to be completed.
  The Manual Assessment of Respiratory Motion (MARM) will be used to assess thoracic and diaphragmatic movements during breathing and quantify their contribution as a percentage of the total breathing movement. During this evaluation, the examiner will position their open hands between posterior and lateral lower rib cage (lower four to six ribs) and the thumbs will vertically be positioned about 1 inch from the spine. In this position, it is possible for the examiner to identify lateral and vertical movements during breathing, as well as upper or lower rib cage predominance. The examiner will draw an upper, lower and horizontal lines starting from the centre of a circle, building a pie chart with the degree of expansion (Courtney et al. 2008, Courtney and van Dixhoorn 2014). A perfect balance between thoracic and abdominal motion during breathing presents a MARM between 0 and 6; as well as a value above 30 may be considered as dysfunctional (Courtney et al. 2011; Courtney et al. 2008).
Breath-holding time | This assessment will be applied only once and takes about 20 minutes to be completed.
  In the Breath-hold test, the variable considered is the total time the participant is able to hold a breath after a normal exhalation at functional residual capacity. This standardized protocol used in participants with DB is called the Buteyko Method of the Control Pause, where the breath is held and timed until the first involuntary motion of the respiratory muscles (Courtney and Cohen 2008). The breath-holding time has been estimated to be approximately 20 seconds patients with DB, while in healthy people is approximately 60 seconds (Jack et al. 2004, Courtney and Cohen 2008). Three attempts will be undertaken with 5-minute rest in between; a stopwatch will be used to time each one, as well as the intervals. The mean of the three attempts will be analysed, in order to remove any learnt effect (Courtney, Greenwood, et al. 2011).

SECONDARY OUTCOMES:
Medical History | This assessment will be applied during the 3-hour assessment, and takes about 5 minutes to be completed.
  Participants will be asked about their medical history, health conditions, comorbidities, medicines in use and its doses.
Age | This assessment will be applied during the 3-hour assessment, and takes about 20 seconds to be completed.
  The date of birth (age) of the participants will be recorded and used for analyses.
Gender | This assessment will be applied during the 3-hour assessment, and takes about 10 seconds to be completed.
  The gender of the participants will be recorded and used for analyses.
Weight | This assessment will be applied during the 3-hour assessment, and takes about 10 seconds to be completed.
  The weight of the participants will be recorded based on self-report.
Height | This assessment will be applied during the 3-hour assessment, and takes about 10 seconds to be completed.
  The height of the participants will be recorded based on self-report.
Body mass index (BMI) | The BMI will be calculated based on height and weight collected from the participants, and will take about 1 minute to be calculated.
  The body mass index of the participants will be calculated as follows: weight over height squared.
Level of physical activity | This assessment will be applied during the 3-hour assessment, and takes about 3 minutes to be completed.
  The level of physical activity of the participants will be recorded based on self-report. They will be asked how many days of a typical week they participate in moderate-to-vigorous physical activity. Also, they will be asked how many minutes per day, during a typical week, they participate in moderate-to-vigorous physical activity. Finally, participants will be asked about any sports that they have participated in and at what level.
Forced vital capacity (FVC) | This assessment will be applied during the 3-hour assessment, and takes about 10 minutes to be completed.
  Lung function will be assessed by spirometry, as hypocapnia is associated with bronchoconstriction (Combes and Fauvage 1997, Brijker et al. 2001). Forced vital capacity (FVC) will be assessed following international recommendations (Miller et al. 2005) and the reference values will be calculated according to Quanjer et al. (1993) and Stanojevic et al. (2010). The participant will be instructed to exhale the maximum possible until residual volume and to inspire as rapid as possible, aiming a maximal and quick gasp until at least 50% of vital capacity.
Forced expiratory volume in the first second (FEV1) | This assessment will be applied during the 3-hour assessment, and takes about 10 minutes to be completed.
  Lung function will be assessed by spirometry, as hypocapnia is associated with bronchoconstriction (Combes and Fauvage 1997, Brijker et al. 2001). Forced expiratory volume in the first second (FEV1) will be assessed following international recommendations (Miller et al. 2005) and the reference values will be calculated according to Quanjer et al. (1993) and Stanojevic et al. (2010). The participant will be instructed to exhale the maximum possible until residual volume and to inspire as rapid as possible, aiming a maximal and quick gasp until at least 50% of vital capacity.
Maximum voluntary ventilation (MVV) | This assessment will be applied during the 3-hour assessment, and takes about 10 minutes to be completed.
  Lung function will be assessed by spirometry, as hypocapnia is associated with bronchoconstriction (Combes and Fauvage 1997, Brijker et al. 2001). Forced expiratory volume in the first second (FEV1) will be assessed following international recommendations (Miller et al. 2005) and the reference values will be calculated according to Quanjer et al. (1993) and Stanojevic et al. (2010). The participant will be instructed to ventilate with her or his maximal ventilation volume and frequency, inhaling and exhaling as deep and quick as possible.
Peak inspiratory flow rate | This assessment will be applied during the 3-hour assessment, and takes about 10 minutes to be completed (together with the FVC, since this outcome is provided by the same manoeuvre).
  The peak inspiratory flow rate will be measured based on the protocol described by McConnell (McConnell 2013). The participant will be instructed to exhale the maximum possible until residual volume and to inspire as rapid as possible, aiming a maximal and quick gasp until at least 50% of vital capacity.
Peak expiratory flow rate | This assessment will be applied during the 3-hour assessment, and takes about 10 minutes to be completed.
  The peak expiratory flow rate will be measured based on the protocol described by McConnell (McConnell 2013). The participant will be instructed to inhale the maximum possible until total vital capacity and to expire as rapid as possible, aiming a maximal and quick manoeuvre.
Inspiratory muscle function | This assessment will be applied during the 3-hour assessment, and takes about 30 minutes to be completed.
  Inspiratory muscle strength will be assessed by the maximal inspiratory pressure (MIP) measurement (McConnell and Copestake 1999, Volianitis et al. 2001) using a mouth pressure meter (Micro Medical RPM, Carefusion, San Diego, United States). The protocol to assess inspiratory muscle strength will be the one described by Black and Hyatt (1969), in which MIP is measured starting at residual volume (McConnell 2013). During the manoeuvre the participants will be instructed to sustain a maximal effort for at least 1.5-2.0 seconds, and a minimum of 5 satisfactory efforts will be considered according to Volianitis et al. (2001).
Expiratory muscle function | This assessment will be applied during the 3-hour assessment, and takes about 30 minutes to be completed.
  Expiratory muscle strength will be assessed by the maximal expiratory pressure (MEP) measurement (McConnell and Copestake 1999, Volianitis et al. 2001) using a mouth pressure meter (Micro Medical RPM, Carefusion, San Diego, United States). The protocol to assess expiratory muscle strength will be the one described by Black and Hyatt (1969), in which MEP is measured starting at total lung capacity (McConnell 2013). During the manoeuvre the participants will be instructed to sustain a maximal effort for at least 1.5-2.0 seconds, and a minimum of 5 satisfactory efforts will be considered according to Volianitis et al. (2001).
Exercise capacity | This assessment will be applied during the 3-hour assessment, and takes about 16 minutes to be completed (simultaneously with the levels of heart rate variability, arterial blood pressure and gas exchange).
  The Astrand-Ryhming submaximal test (Astrand and Ryhming 1954) will be used to assess exercise capacity of all participants and to predict maximal oxygen uptake. Participants will be instructed to stay 48 hours previous to the test without practicing exercise. This test will be performed on a cycle ergometer and power outputs of 75 to 150 watts and 100 to 200 watts will be used for women and men, respectively. The rotation of 50 rpm needs to be kept for 6 minutes. The HR is registered at the 5th and 6th minutes of the exercise test, and with the right load, these values cannot differentiate from each other more than 5 bpm. After that, a mathematic model will be used to predict the maximal oxygen uptake (Astrand and Ryhming 1954, Legge and Banister 1986, Macsween 2001).
Level of heart rate variability | This assessment will be applied during the 3-hour assessment, and takes about 15 minutes to be placed and will be continuously used during the exercise test (16 minutes) and the slow-breathing task (15 minutes).
  The heart rate variability (HRV) will be continuously assessed during five minutes before, during, and five minutes after the exercise test and during a controlled breathing of approximately 6-10 breaths per minute. HRV will be assessed by using a Polar® V800 device (Polar, Kempele-Finland), and the heart's electrical signal will be processed by using Kubios HRV version 2.2. The data will be initially filtered and smoothed to obtain heart rate frequency mean, time-domain analyses of the R-R intervals (interval between 2 "R" curves in the electrocardiogram (e.g., standard deviation of normal-to-normal RR intervals [SDNN] and root mean square of successive differences [RMSSD]) and spectral analyses of frequency indices (i.e., very low-frequency [0-0.04], low-frequency [0.04-0.15 Hz] and high-frequency [0.15-0.4 Hz]) aiming the further understanding of the autonomic nervous system responses in DB.
Level of arterial blood pressure | This assessment will be applied during the 3-hour assessment, and takes about 15 minutes to be placed and will be continuously used during the exercise test (16 minutes) and the slow-breathing task (15 minutes).
  The arterial blood pressure (ABP) will be continuously assessed during five minutes before, during, and five minutes after the exercise test and during a controlled breathing of approximately 6-10 breaths per minute. Finger ABP will be measured by the use of Finometer 1.10 (Finapres Medical System, Amsterdam - The Netherlands), which non-invasively registers continuous blood pressure measurements. The finger pressure generates a waveform and the ABP is exported based on calculations built every heartbeat (Bogert and van Lieshout 2005). Finger ABP signals will be processed by using the Lab Chart Pro Software, which records, displays and analyses real time data from up to 32 channels.
Minute volume | This assessment will be applied during the 3-hour assessment, and takes about 15 minutes to be placed and will be continuously used during the exercise test (16 minutes) and the slow-breathing task (15 minutes).
  The indirect calorimetry (IC) will be performed by the portable system K5® (Cosmed, Rome, Italy). This ergospirometer calculates breath-by-breath oscillations of minute volume (VE). The device will be attached to the participant's chest and a facemask, which has less than 30 ml of dead space, suitably adjusted to eliminate air leakage. The equipment will be programmed to assess data breath-by-breath and an average will be recorded every 5 seconds. Oxycon Pro software will be used to process the data for further analyses.
Oxygen Uptake | This assessment will be applied during the 3-hour assessment, and takes about 15 minutes to be placed and will be continuously used during the exercise test (16 minutes) and the slow-breathing task (15 minutes).
  The indirect calorimetry (IC) will be performed by the portable system K5® (Cosmed, Rome, Italy). This ergospirometer calculates breath-by-breath oscillations of oxygen uptake (O2). The device will be attached to the participant's chest and a facemask, which has less than 30 ml of dead space, suitably adjusted to eliminate air leakage. The equipment will be programmed to assess data breath-by-breath and an average will be recorded every 5 seconds. Oxycon Pro software will be used to process the data for further analyses.
Carbon dioxide | This assessment will be applied during the 3-hour assessment, and takes about 15 minutes to be placed and will be continuously used during the exercise test (16 minutes) and the slow-breathing task (15 minutes).
  The indirect calorimetry (IC) will be performed by the portable system K5® (Cosmed, Rome, Italy). This ergospirometer calculates breath-by-breath oscillations of carbon dioxide (CO2). The device will be attached to the participant's chest and a facemask, which has less than 30 ml of dead space, suitably adjusted to eliminate air leakage. The equipment will be programmed to assess data breath-by-breath and an average will be recorded every 5 seconds. Oxycon Pro software will be used to process the data for further analyses.
Respiratory exchange ratio | This assessment will be applied during the 3-hour assessment, and takes about 15 minutes to be placed and will be continuously used during the exercise test (16 minutes) and the slow-breathing task (15 minutes).
  The indirect calorimetry (IC) will be performed by the portable system K5® (Cosmed, Rome, Italy). This ergospirometer calculates breath-by-breath oscillations of respiratory exchange ratio (RER). The device will be attached to the participant's chest and a facemask, which has less than 30 ml of dead space, suitably adjusted to eliminate air leakage. The equipment will be programmed to assess data breath-by-breath and an average will be recorded every 5 seconds. Oxycon Pro software will be used to process the data for further analyses.
Respiratory rate | This assessment will be applied during the 3-hour assessment, and takes about 15 minutes to be placed and will be continuously used during the exercise test (16 minutes) and the slow-breathing task (15 minutes).
  The indirect calorimetry (IC) will be performed by the portable system K5® (Cosmed, Rome, Italy). This ergospirometer calculates breath-by-breath oscillations of respiratory rate (breaths per minute - BPM). The device will be attached to the participant's chest and a facemask, which has less than 30 ml of dead space, suitably adjusted to eliminate air leakage. The equipment will be programmed to assess data breath-by-breath and an average will be recorded every 5 seconds. Oxycon Pro software will be used to process the data for further analyses.
Attentional focus | This assessment will be applied 3 times during the exercise test, and takes about 30 seconds to be completed each time. So, it will take approximately 1 minute and 30 seconds to be applied in total.
  Attentional focus (Attention Scale [AS]; Tammen 1996, Tenenbaum et al. 2007) will be measured at various time points (pre exercise, at the 3rd minute, and at the end of the exercise test) during the execution of the six-minute cycling test described above.
Level of fatigue | This assessment will be applied 3 times during the exercise test, and takes about 15 seconds to be completed each time. So, it will take approximately 45 seconds to be applied in total.
  Limb discomfort (Category Ratio 10 [CR10-fatigue]; Borg 1982) (Borg Scale fatigue) will be measured at various time points (pre exercise, at the 3rd minute, and at the end of the exercise test) during the execution of the six-minute cycling test described above.
Level of dyspnoea | This assessment will be applied 3 times during the exercise test, and takes about 15 seconds to be completed each time. So, it will take approximately 45 seconds to be applied in total.
  Dyspnoea (CR10-dyspnoea; Borg 1982) (Borg Scale dyspnoea) will be measured at various time points (pre exercise, at the 3rd minute, and at the end of the exercise test) during the execution of the six-minute cycling test described above.

CONTACTS AND LOCATIONS:
Overall Officials: Panagiota Smyrni, Dr, Study Chair — Brunel University London
Locations (1):
- Brunel University London, London, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barker N, Everard ML. Getting to grips with 'dysfunctional breathing'. Paediatr Respir Rev. 2015 Jan;16(1):53-61. doi: 10.1016/j.prrv.2014.10.001. Epub 2014 Nov 25. PMID 25499573
- [Background] Barker NJ, Jones M, O'Connell NE, Everard ML. Breathing exercises for dysfunctional breathing/hyperventilation syndrome in children. Cochrane Database Syst Rev. 2013 Dec 18;2013(12):CD010376. doi: 10.1002/14651858.CD010376.pub2. PMID 24347088
- [Background] Bott J, Blumenthal S, Buxton M, Ellum S, Falconer C, Garrod R, Harvey A, Hughes T, Lincoln M, Mikelsons C, Potter C, Pryor J, Rimington L, Sinfield F, Thompson C, Vaughn P, White J; British Thoracic Society Physiotherapy Guideline Development Group. Guidelines for the physiotherapy management of the adult, medical, spontaneously breathing patient. Thorax. 2009 May;64 Suppl 1:i1-51. doi: 10.1136/thx.2008.110726. No abstract available. PMID 19406863
- [Background] Brashear RE. Hyperventilation syndrome. Lung. 1983;161(5):257-73. doi: 10.1007/BF02713872. No abstract available. PMID 6138480
- [Background] Courtney R, Greenwood KM, Cohen M. Relationships between measures of dysfunctional breathing in a population with concerns about their breathing. J Bodyw Mov Ther. 2011 Jan;15(1):24-34. doi: 10.1016/j.jbmt.2010.06.004. Epub 2010 Jul 16. PMID 21147415
- [Background] Gridina I, Bidat E, Chevallier B, Stheneur C. [Prevalence of chronic hyperventilation syndrome in children and teenagers]. Arch Pediatr. 2013 Mar;20(3):265-8. doi: 10.1016/j.arcped.2012.12.016. Epub 2013 Feb 1. French. PMID 23375424
- [Background] de Groot EP, Duiverman EJ, Brand PL. Dysfunctional breathing in children with asthma: a rare but relevant comorbidity. Eur Respir J. 2013 May;41(5):1068-73. doi: 10.1183/09031936.00130212. Epub 2012 Sep 27. PMID 23018913
- [Background] Hagman C, Janson C, Emtner M. A comparison between patients with dysfunctional breathing and patients with asthma. Clin Respir J. 2008 Apr;2(2):86-91. doi: 10.1111/j.1752-699X.2007.00036.x. PMID 20298312
- [Background] Hagman C, Janson C, Emtner M. Breathing retraining - a five-year follow-up of patients with dysfunctional breathing. Respir Med. 2011 Aug;105(8):1153-9. doi: 10.1016/j.rmed.2011.03.006. Epub 2011 Mar 31. PMID 21454062
- [Background] Howell JB. The hyperventilation syndrome: a syndrome under threat? Thorax. 1997 Aug;52 Suppl 3(Suppl 3):S30-4. doi: 10.1136/thx.52.2008.s30. No abstract available. PMID 9381424
- [Background] Jones M, Harvey A, Marston L, O'Connell NE. Breathing exercises for dysfunctional breathing/hyperventilation syndrome in adults. Cochrane Database Syst Rev. 2013 May 31;2013(5):CD009041. doi: 10.1002/14651858.CD009041.pub2. PMID 23728685
- [Background] Jones M, Troup F, Nugus J, Roughton M, Hodson M, Rayner C, Bowen F, Pryor J. Does manual therapy provide additional benefit to breathing retraining in the management of dysfunctional breathing? A randomised controlled trial. Disabil Rehabil. 2015;37(9):763-70. doi: 10.3109/09638288.2014.941020. Epub 2014 Jul 15. PMID 25026508
- [Background] LEWIS BI. Hyperventilation syndrome: a clinical and physiological evaluation. Calif Med. 1959 Sep;91(3):121-6. PMID 14416492
- [Background] Magarian GJ. Hyperventilation syndromes: infrequently recognized common expressions of anxiety and stress. Medicine (Baltimore). 1982 Jul;61(4):219-36. No abstract available. PMID 7045570
- [Background] Morgan MD. Dysfunctional breathing in asthma: is it common, identifiable and correctable? Thorax. 2002 Oct;57 Suppl 2(Suppl 2):II31-II35. No abstract available. PMID 12364708
- [Background] Peroni DG, Piacentini GL, Bodini A, Boner AL. Childhood Asthma Control Test in asthmatic children with dysfunctional breathing. J Allergy Clin Immunol. 2008 Jan;121(1):266-7; author reply 267. doi: 10.1016/j.jaci.2007.06.049. Epub 2007 Oct 17. No abstract available. PMID 17920668
- [Background] Thomas M, McKinley RK, Freeman E, Foy C. Prevalence of dysfunctional breathing in patients treated for asthma in primary care: cross sectional survey. BMJ. 2001 May 5;322(7294):1098-100. doi: 10.1136/bmj.322.7294.1098. PMID 11337441
- [Background] Thomas M, McKinley RK, Freeman E, Foy C, Price D. The prevalence of dysfunctional breathing in adults in the community with and without asthma. Prim Care Respir J. 2005 Apr;14(2):78-82. doi: 10.1016/j.pcrj.2004.10.007. PMID 16701702
- [Background] van Dixhoorn J, Duivenvoorden HJ. Efficacy of Nijmegen Questionnaire in recognition of the hyperventilation syndrome. J Psychosom Res. 1985;29(2):199-206. doi: 10.1016/0022-3999(85)90042-x. PMID 4009520
- [Background] van Dixhoorn J, Folgering H. The Nijmegen Questionnaire and dysfunctional breathing. ERJ Open Res. 2015 May 15;1(1):00001-2015. doi: 10.1183/23120541.00001-2015. eCollection 2015 May. PMID 27730128
- [Background] Vansteenkiste J, Rochette F, Demedts M. Diagnostic tests of hyperventilation syndrome. Eur Respir J. 1991 Apr;4(4):393-9. PMID 1855568
- [Background] Aadland E, Ylvisaker E. Reliability of the Actigraph GT3X+ Accelerometer in Adults under Free-Living Conditions. PLoS One. 2015 Aug 14;10(8):e0134606. doi: 10.1371/journal.pone.0134606. eCollection 2015. PMID 26274586
- [Background] ASTRAND PO, RYHMING I. A nomogram for calculation of aerobic capacity (physical fitness) from pulse rate during sub-maximal work. J Appl Physiol. 1954 Sep;7(2):218-21. doi: 10.1152/jappl.1954.7.2.218. No abstract available. PMID 13211501
- [Background] Bernardi L, Porta C, Gabutti A, Spicuzza L, Sleight P. Modulatory effects of respiration. Auton Neurosci. 2001 Jul 20;90(1-2):47-56. doi: 10.1016/S1566-0702(01)00267-3. PMID 11485292
- [Background] Bernardi L, Wdowczyk-Szulc J, Valenti C, Castoldi S, Passino C, Spadacini G, Sleight P. Effects of controlled breathing, mental activity and mental stress with or without verbalization on heart rate variability. J Am Coll Cardiol. 2000 May;35(6):1462-9. doi: 10.1016/s0735-1097(00)00595-7. PMID 10807448
- [Background] Bjelland I, Dahl AA, Haug TT, Neckelmann D. The validity of the Hospital Anxiety and Depression Scale. An updated literature review. J Psychosom Res. 2002 Feb;52(2):69-77. doi: 10.1016/s0022-3999(01)00296-3. PMID 11832252
- [Background] Bogert LW, van Lieshout JJ. Non-invasive pulsatile arterial pressure and stroke volume changes from the human finger. Exp Physiol. 2005 Jul;90(4):437-46. doi: 10.1113/expphysiol.2005.030262. Epub 2005 Mar 31. PMID 15802289
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Background] Brijker F, van den Elshout FJ, Heijdra YF, Bosch FH, Folgering HT. Effect of acute metabolic acid/base shifts on the human airway calibre. Respir Physiol. 2001 Jan;124(2):151-8. doi: 10.1016/s0034-5687(00)00196-1. PMID 11164206
- [Background] Combes P, Fauvage B. Combined effects of hypocapnia and nicardipine on airway resistance: a pilot study. Eur J Clin Pharmacol. 1997;51(5):385-8. doi: 10.1007/s002280050218. PMID 9049579
- [Background] Courtney R, Cohen M. Investigating the claims of Konstantin Buteyko, M.D., Ph.D.: the relationship of breath holding time to end tidal CO2 and other proposed measures of dysfunctional breathing. J Altern Complement Med. 2008 Mar;14(2):115-23. doi: 10.1089/acm.2007.7204. PMID 18315509
- [Background] Courtney R, van Dixhoorn J, Cohen M. Evaluation of breathing pattern: comparison of a Manual Assessment of Respiratory Motion (MARM) and respiratory induction plethysmography. Appl Psychophysiol Biofeedback. 2008 Jun;33(2):91-100. doi: 10.1007/s10484-008-9052-3. Epub 2008 Mar 5. PMID 18320303
- [Background] Courtney R, van Dixhoorn J, Greenwood KM, Anthonissen EL. Medically unexplained dyspnea: partly moderated by dysfunctional (thoracic dominant) breathing pattern. J Asthma. 2011 Apr;48(3):259-65. doi: 10.3109/02770903.2011.554942. Epub 2011 Feb 22. PMID 21341969
- [Background] Guelen I, Westerhof BE, Van Der Sar GL, Van Montfrans GA, Kiemeneij F, Wesseling KH, Bos WJ. Finometer, finger pressure measurements with the possibility to reconstruct brachial pressure. Blood Press Monit. 2003 Feb;8(1):27-30. doi: 10.1097/00126097-200302000-00006. PMID 12604933
- [Background] Han JN, Stegen K, Simkens K, Cauberghs M, Schepers R, Van den Bergh O, Clement J, Van de Woestijne KP. Unsteadiness of breathing in patients with hyperventilation syndrome and anxiety disorders. Eur Respir J. 1997 Jan;10(1):167-76. doi: 10.1183/09031936.97.10010167. PMID 9032511
- [Background] Hawkes EZ, Nowicky AV, McConnell AK. Diaphragm and intercostal surface EMG and muscle performance after acute inspiratory muscle loading. Respir Physiol Neurobiol. 2007 Mar 15;155(3):213-9. doi: 10.1016/j.resp.2006.06.002. Epub 2006 Jul 18. PMID 16846758
- [Background] Healy GN, Clark BK, Winkler EA, Gardiner PA, Brown WJ, Matthews CE. Measurement of adults' sedentary time in population-based studies. Am J Prev Med. 2011 Aug;41(2):216-27. doi: 10.1016/j.amepre.2011.05.005. PMID 21767730
- [Background] Homma I, Masaoka Y. Breathing rhythms and emotions. Exp Physiol. 2008 Sep;93(9):1011-21. doi: 10.1113/expphysiol.2008.042424. Epub 2008 May 16. PMID 18487316
- [Background] Imholz BP, Wieling W, van Montfrans GA, Wesseling KH. Fifteen years experience with finger arterial pressure monitoring: assessment of the technology. Cardiovasc Res. 1998 Jun;38(3):605-16. doi: 10.1016/s0008-6363(98)00067-4. PMID 9747429
- [Background] Jack S, Rossiter HB, Pearson MG, Ward SA, Warburton CJ, Whipp BJ. Ventilatory responses to inhaled carbon dioxide, hypoxia, and exercise in idiopathic hyperventilation. Am J Respir Crit Care Med. 2004 Jul 15;170(2):118-25. doi: 10.1164/rccm.200207-720OC. Epub 2004 Apr 1. PMID 15059786
- [Background] Jenkinson C, Stewart-Brown S, Petersen S, Paice C. Assessment of the SF-36 version 2 in the United Kingdom. J Epidemiol Community Health. 1999 Jan;53(1):46-50. doi: 10.1136/jech.53.1.46. PMID 10326053
- [Background] Joseph CN, Porta C, Casucci G, Casiraghi N, Maffeis M, Rossi M, Bernardi L. Slow breathing improves arterial baroreflex sensitivity and decreases blood pressure in essential hypertension. Hypertension. 2005 Oct;46(4):714-8. doi: 10.1161/01.HYP.0000179581.68566.7d. Epub 2005 Aug 29. PMID 16129818
- [Background] Juniper EF, O'Byrne PM, Guyatt GH, Ferrie PJ, King DR. Development and validation of a questionnaire to measure asthma control. Eur Respir J. 1999 Oct;14(4):902-7. doi: 10.1034/j.1399-3003.1999.14d29.x. PMID 10573240
- [Background] Kozey-Keadle S, Libertine A, Lyden K, Staudenmayer J, Freedson PS. Validation of wearable monitors for assessing sedentary behavior. Med Sci Sports Exerc. 2011 Aug;43(8):1561-7. doi: 10.1249/MSS.0b013e31820ce174. PMID 21233777
- [Background] Legge BJ, Banister EW. The Astrand-Ryhming nomogram revisited. J Appl Physiol (1985). 1986 Sep;61(3):1203-9. doi: 10.1152/jappl.1986.61.3.1203. PMID 3759759
- [Background] Lehrer PM, Vaschillo E, Vaschillo B. Resonant frequency biofeedback training to increase cardiac variability: rationale and manual for training. Appl Psychophysiol Biofeedback. 2000 Sep;25(3):177-91. doi: 10.1023/a:1009554825745. PMID 10999236
- [Background] Lum LC. Hyperventilation and anxiety state. J R Soc Med. 1981 Jan;74(1):1-4. doi: 10.1177/014107688107400101. No abstract available. PMID 6780688
- [Background] Lyden K, Kozey Keadle SL, Staudenmayer JW, Freedson PS. Validity of two wearable monitors to estimate breaks from sedentary time. Med Sci Sports Exerc. 2012 Nov;44(11):2243-52. doi: 10.1249/MSS.0b013e318260c477. PMID 22648343
- [Background] Macsween A. The reliability and validity of the Astrand nomogram and linear extrapolation for deriving VO2max from submaximal exercise data. J Sports Med Phys Fitness. 2001 Sep;41(3):312-7. PMID 11533560
- [Background] Matthews CE, Chen KY, Freedson PS, Buchowski MS, Beech BM, Pate RR, Troiano RP. Amount of time spent in sedentary behaviors in the United States, 2003-2004. Am J Epidemiol. 2008 Apr 1;167(7):875-81. doi: 10.1093/aje/kwm390. Epub 2008 Feb 25. PMID 18303006
- [Background] McConnell AK, Copestake AJ. Maximum static respiratory pressures in healthy elderly men and women: issues of reproducibility and interpretation. Respiration. 1999;66(3):251-8. doi: 10.1159/000029386. PMID 10364742
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Background] Mitchell AJ, Bacon CJ, Moran RW. Reliability and Determinants of Self-Evaluation of Breathing Questionnaire (SEBQ) Score: A Symptoms-Based Measure of Dysfunctional Breathing. Appl Psychophysiol Biofeedback. 2016 Mar;41(1):111-20. doi: 10.1007/s10484-015-9316-7. PMID 26400252
- [Background] Murias JM, Kowalchuk JM, Paterson DH. Speeding of VO2 kinetics with endurance training in old and young men is associated with improved matching of local O2 delivery to muscle O2 utilization. J Appl Physiol (1985). 2010 Apr;108(4):913-22. doi: 10.1152/japplphysiol.01355.2009. Epub 2010 Feb 11. PMID 20150562
- [Background] Quanjer PH, Tammeling GJ, Cotes JE, Pedersen OF, Peslin R, Yernault JC. Lung volumes and forced ventilatory flows. Report Working Party Standardization of Lung Function Tests, European Community for Steel and Coal. Official Statement of the European Respiratory Society. Eur Respir J Suppl. 1993 Mar;16:5-40. No abstract available. PMID 8499054
- [Background] RAHN H, OTIS AB, et al. The pressure-volume diagram of the thorax and lung. Am J Physiol. 1946;146(2):161-78. doi: 10.1152/ajplegacy.1946.146.2.161. No abstract available. PMID 20982947
- [Background] Sclauser Pessoa IM, Franco Parreira V, Fregonezi GA, Sheel AW, Chung F, Reid WD. Reference values for maximal inspiratory pressure: a systematic review. Can Respir J. 2014 Jan-Feb;21(1):43-50. doi: 10.1155/2014/982374. Epub 2013 Oct 17. PMID 24137574
- [Background] Stanojevic S, Wade A, Stocks J. Reference values for lung function: past, present and future. Eur Respir J. 2010 Jul;36(1):12-9. doi: 10.1183/09031936.00143209. PMID 20595163
- [Background] Volianitis S, McConnell AK, Jones DA. Assessment of maximum inspiratory pressure. Prior submaximal respiratory muscle activity ('warm-up') enhances maximum inspiratory activity and attenuates the learning effect of repeated measurement. Respiration. 2001;68(1):22-7. doi: 10.1159/000050458. PMID 11223726
- [Background] Warburton CJ, Jack S. Can you diagnose hyperventilation? Chron Respir Dis. 2006;3(3):113-5. doi: 10.1191/1479972306cd116ed. No abstract available. PMID 16916004
- [Background] Ware JE Jr. SF-36 health survey update. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3130-9. doi: 10.1097/00007632-200012150-00008. No abstract available. PMID 11124729
- [Background] Ware JE Jr, Gandek B. Overview of the SF-36 Health Survey and the International Quality of Life Assessment (IQOLA) Project. J Clin Epidemiol. 1998 Nov;51(11):903-12. doi: 10.1016/s0895-4356(98)00081-x. PMID 9817107
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820